CLINICAL TRIAL: NCT01473927
Title: Significance of Ficolin 2 in the Determination of Serological Activity in Chronic Inflammatory Bowel Disease
Status: Completed | Type: Observational
Sponsor: University of Bern (Other)
Collaborators: University Hospital, Basel, Switzerland (Other); University of Lausanne Hospitals (Other); Swiss IBD Cohort Study (Unknown); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Seibold Prof. Dr. med., Spital Tiefenau Bern / Inselspital Bern
Other Study IDs: 110/06
Record Dates: First submitted 2011-11-03; First posted 2011-11-17 (Estimated); Last update posted 2014-03-12 (Estimated); Status verified 2014-03

CONDITIONS: Crohn Disease
Keywords: Inflammatory bowel diseases; Crohn disease; Ficolin-2; C-Reactive Protein; Calprotectin; Inflammatory markers; SES-CD
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases | interventions — Endoscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Serum Stool
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Crohn's Disease patients
  Interventions: Other: Endoscopy
- 2: Ulcerative colitis patients
  Interventions: Other: Endoscopy

INTERVENTIONS:
Other: Endoscopy — Only patients undergoing endoscopy for clinical reasons will be included in the study, i.e. no endoscopies will be performed solely for study reasons. For the purposes of our study, endoscopy serves to determine the degree of inflammation and no additional biopsies are taken. Blood for CRP and ficolin-2 analysis will be taken through the Venflon® installed for endoscopy.
  Groups: 1
Other: Endoscopy — Only patients undergoing endoscopy for clinical reasons will be included in the study, i.e. no endoscopies will be performed solely for study reasons. For the purposes of our study, endoscopy serves to determine the degree of inflammation and no additional biopsies are taken. Blood for CRP and ficolin-2 analysis will be taken through the Venflon® installed for endoscopy.
  Groups: 2

SUMMARY:
Background Determining disease activity in IBD is sometimes difficult and, to be accurate, requires endoscopy. The serum marker CRP has not proven sufficiently valuable as a marker for IBD specific inflammation. As an alternative, so far fecal calprotectin appears to be more reliable and has shown a certain value as predictive marker. Our preliminary data now show, that the serum concentrations of ficolin-2 are significantly higher in CD patients with a HBI >3. Ficolin-2 is a lectin and acute phase protein produced in the liver and, like MBL, can activate the lectin pathway of complement. Unlike MBL, deficiency for ficolin-2 was not detected in our patient cohort, nor could we find functional deficiencies for ficolin-2 (paper submitted).

Study Aims The study is aimed to substantiate the data from our pilot study which shows that ficolin-2 is significantly increased in CD patients during inflammation. Therefore, the study will measure ficolin-2 concentrations in a sufficiently large patient group to obtain enough statistical power and to compare these results with the endoscopic disease score (SES-CD) and CRP and calprotectin values. Statistical analysis of the data will show us if ficolin-2 is a reliable and easy to obtain new marker for active inflammation in CD.

Study Design Based on a power analysis 112 CD patients and 112 UC patients need to be analyzed. They will be recruited from Bern, Basel and Lausanne. Only patients with routine endoscopy will be included in the study and will be scored by SES-CD. Blood samples will be collected at the day of endoscopy. Stool sample will be collected within the same week of endoscopy. Calprotectin and CRP concentrations will be determined by routine diagnostics, ficolin-2 concentrations will be determined by ELISA in our laboratory. Finally, all data will be statistically analyzed.

DETAILED DESCRIPTION:
Background

Background Like mannan-binding lectin (MBL), ficolins are important soluble receptors for microbial associated molecular patterns leading to the activation of the lectin pathway complement. Ficolins are structurally related to MBL, but due to their different carbohydrate recognition domain represent an own family of lectins (1). The single polypeptide chains of ficolins form trimers and the trimers finally form higher order structures (tetramers up to hexamers) which constitute the functional protein. Humans have three ficolins: Ficolin-1 (M-ficolin), -2 (L-ficolin) and -3 (H-ficolin), whereas ficolin-2 and -3 are present in the serum, ficolin-1 is found on the surface of monocytes. Both, ficolin-2 and -3 are produced in the liver with an additional source for ficolin-3 in the lung. Like MBL, ficolins have to assemble with the MBL-associated serin proteases (MASPs) in order to activate the complement pathway (1). In our study on a possible role for the influence of the complement system in the development of CD-associated anti-Saccharomyces cerevisiae antibodies (ASCAs), we noticed that chronic inflammatory bowel disease (CIBD) patients, specifically Crohn's disease (CD) patients, exhibited high serum ficolin 2 concentrations.

Our research group is interested in the interaction of the innate immune system with microorganisms of the intestinal flora, focusing on possible defects in innate immune mechanisms. We have more than ten years experience in the field, with a special focus on ASCA and MBL. We have been able to continuously publish our work about these theories.

Our earlier and present studies on the role of MBL and the lectin pathway of complement in CD led to the finding of increased ficolin-2 concentration in the sera of CD patients. Moreover, we found that CD patients with a Harvey-Bradshaw index >3 had significantly higher ficolin 2 concentrations than those with a Harvey-Bradshaw index of ≤ 3.

Study Hypotheses

The following hypotheses are to be tested:

1. The ficolin 2 concentration is higher in Crohn's patients with active disease than in CD patients in remission.
2. Ficolin 2 correlates with endoscopic activity.
3. Ficolin 2 correlates with calprotectin.

Objective

The findings from the first part of the study are to be confirmed in a prospective and more detailed study with a larger patient cohort, testing our (new) working hypothesis that ficolin 2 represents a serum marker for disease activity in CD.

Since it is currently difficult to reliably determine disease activity in CD patients using serum and stool markers without simultaneous endoscopic examination, another specific and easy to obtain disease marker which correlates well with disease activity would be highly welcome. Particularly because the current standard marker, to monitor disease activity (faecal calprotectin), is much less accepted than testing for parameters in the blood.

Therefore, the study aims at answering the question of whether ficolin 2 is present in greater concentrations in the blood of Crohn's patients with active inflammation compared to CD patients in remission or to ulcerative colitis (UC) patients.

Methods

For the purposes of the study, the endoscopic activity index will be recorded using the SES-CD (simplified endoscopic score for CD) for Crohn's patients and the Mayo score for colitis patients.

Approximately 5 ml blood will be taken to prepare serum. (5.5 ml or 4.9 ml S Monovette or 4.7 ml or 4.9 ml serum gel Monovette).

A second test tube of blood will be taken for CRP determination. In order to measure calprotectin, the patient will be asked to provide a stool sample shortly before or shortly after the endoscopic examination (within one week).

Serum ficolin values are measured by enzyme-linked immune sorbent assay (ELISA) in the laboratory at the Department of Clinical Research, University of Bern; all other values are determined in routine diagnostic laboratories.

ELIGIBILITY:
Inclusion Criteria:

* known IBD
* endoscopy for clinical reasons
* enrolled in the Swiss IBD cohort study

Exclusion Criteria

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All CD and UC patients undergoing endoscopy for clinical reasons at one of the involved clinical centers.
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2011-10; Primary Completion 2013-02 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Ficolin-2 concentration in serum | During endoscopy

SECONDARY OUTCOMES:
CRP concentration in serum | During endoscopy
Calprotectin in stool sample | One week before endoscopy up to one week after endoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Frank Seibold, Prof. Dr. med., Study Director — Spital Tiefenau / Inselspital Bern
Locations (3):
- Switzerland (3):
  - Gastroenterology and Hepatology, Basel University Hospital, Basel, Canton of Basel-City
  - DCR, Gastroenterology, Bern, University of Bern, Bern, Canton of Bern
  - Service de gastro-entérologie et hépatologie, CHUV Lausanne, Lausanne, Canton of Vaud

REFERENCES:
- [Background] Holmskov U, Thiel S, Jensenius JC. Collections and ficolins: humoral lectins of the innate immune defense. Annu Rev Immunol. 2003;21:547-78. doi: 10.1146/annurev.immunol.21.120601.140954. Epub 2001 Dec 19. PMID 12524383